CLINICAL TRIAL: NCT04098809
Title: Impact of Catheter Size on Peri-Operative Pain After Robotic Assisted Laparoscopic Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benaroya Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB17-095
Record Dates: First submitted 2019-09-11; First posted 2019-09-23 (Actual); Results first posted 2019-12-26 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Catheter 16 French (Active Comparator): 16 French urinary catheter
  Interventions: Device: 16 French urinary catheter
- Catheter 20 French (Active Comparator): 20 French urinary catheter
  Interventions: Device: 20 French urinary catheter

INTERVENTIONS:
Device: 16 French urinary catheter — 16 French urinary catheter
  Arms: Catheter 16 French
Device: 20 French urinary catheter — 20 French urinary catheter
  Arms: Catheter 20 French

SUMMARY:
This study is designed to assess the effect of catheter size on postoperative catheter pain, urinary continence, urinary flow rates, post void residuals, International Prostate Symptom Scores (IPSS), and Quality of Life (QoL) score, as well as long term complications after robotic assisted laparoscopic prostatectomy.

DETAILED DESCRIPTION:
Subjects identified to receive a robotic assisted laparoscopic prostatectomy.were randomized to either a 16 French or 20 French catheter at the completion of the prostatectomy. All prostatectomies were performed by one of three surgeons at the investigator's institution. Preoperative demographics and operative data were recorded for each group. Catheters remained in place for 7-14 days. Subjects were asked on postoperative day 7 to report their catheter-related pain and amount of opioid medication used. Urinary symptoms and quality of life scores and pads per day were recorded at 6 weeks and 12 weeks post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Identified as candidate for robotic assisted laparoscopic prostatectomy

Exclusion Criteria:

* Having filled a prescription for opioid medication in last 2 months.
* Known latex allergy
* Known pre-operatively that catheter placement will exceed 14 days
* History of pelvic radiation
* Significant deviation from normal operative protocol

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2018-11-07 (Actual); Study Completion 2018-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Corman, MD, Principal Investigator — Virginia Mason Medical Center
Locations (1):
- Virginia Mason Medical center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Catheter 16 French | Catheter 20 French
Started | 27 | 25
Completed | 24 | 21
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Physician Decision | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Catheter 16 French: 16 French urinary catheter
  Patients will be randomized by chance to either a 16 French or 20 French catheter in a 1:1 ratio.
- Catheter 20 French: 20 French urinary catheter
  Patients will be randomized by chance to either a 16 French or 20 French catheter in a 1:1 ratio.
- Total: Total of all reporting groups
Arm/Group | Catheter 16 French | Catheter 20 French | Total
Number analyzed (Participants) | 24 | 21 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.17 (7.01) | 62.57 (5.95) | 62.89 (6.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 24 | 21 | 45
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.77 (3.25) | 27.02 (3.33) | 27.42 (3.27)
Prior Abdominal Surgery [Count of Participants; unit: Participants]
  Prior Abdominal Surgery - No | 14 | 17 | 31
  Prior Abdominal Surgery - Yes | 10 | 4 | 14
Chronic Pain [Count of Participants; unit: Participants]
  Chronic Pain - No | 23 | 20 | 43
  Chronic Pain - Yes | 1 | 1 | 2
Previous Transurethral Resection of Prostate (TURP) [Count of Participants; unit: Participants]
  Previous TURP - No | 23 | 21 | 44
  Previous TURP -Yes | 1 | 0 | 1
International Prostate Symptom Score [Mean (Standard Deviation); unit: score] — International Prostate Symptom Score allow the urologist to better understand the severity of urinary voiding symptoms. The scale includes 7 questions with a scale range from 1-5.
  The overall range is 0- 35. Higher values represent a worse outcome.
  score | 9.24 (6.09) | 10.00 (5.78) | 9.59 (5.88)
Baseline Quality of Life [Mean (Standard Deviation); unit: Score] — Quality of life, as perceived by the patient, is assessed using the eighth question of the International Prostate Symptom Score. This question asks "If you were to spend the rest of your life with your urinary condition the way it is now, how would you feel about that?" The range is from a score of 1 (delighted) to 6 (terrible) and the lower the score, the better the outcome.
  Score | 1.65 (1.27) | 2.11 (1.18) | 1.89 (1.23)
International Index of Erectile Function [Mean (Standard Deviation); unit: score] — International Index of Erectile Function (IIEF) Questionnaire is a validated, multi-dimensional, self-administered questionnaire that has been found useful in the clinical assessment of erectile dysfunction and treatment outcomes in clinical trials. The range for each of 5 questions 1 9very low) to 5 (very high). The total score can then range from 5 to 25. The higher the score the better the outcome.
  score | 18.85 (6.83) | 17.39 (7.57) | 18.16 (7.13)
TNM Stage [Count of Participants; unit: Participants] — This staging system is a standard method for the cancer care team to describe how far a cancer has spread. The TNM system is based on 5 key pieces of information:the size and extent of the primary Tumor (T category),whether the cancer has spread to nearby lymph Nodes (N Category),the absence or presence of cancer outside the prostate, or metastasis (M Category).
  Participants
    T2N0 | 6 | 4 | 10
    T2NX | 5 | 6 | 11
    T2cN0 | 1 | 1 | 2
    T3aN0 | 9 | 10 | 19
    T3bN0 | 2 | 0 | 2
    T3bN1 | 1 | 0 | 1
Gleason Score [Count of Participants; unit: Participants] — The Prostate Cancer Gleason Score score ranges from 2 to 10. To determine the score, the pathologist uses a microscope to look at the patterns of cells in the prostate tissue. The most common cell pattern is given a grade of 1 (most like normal cells) to 5 (most abnormal).The pathologist will assign one Gleason grade to the most predominant pattern in your biopsy and a second Gleason grade to the second most predominant pattern and then add the 2 numbers together. A Gleason score of 6 is low grade, 7 is intermediate grade, and a score of 8 to 10 is high grade cancer.
  Participants
    Gleason 6 | 7 | 7 | 14
    Gleason 7 | 17 | 13 | 30
    Gleason 8 | 0 | 1 | 1
Extra Prostatic Extension [Count of Participants; unit: Participants]
  Extra Prostatic Extension - No | 12 | 11 | 23
  Extra Prostatic Extension - Yes | 12 | 10 | 22
Seminal Vesical Invasion [Count of Participants; unit: Participants]
  Seminal Vesical Invasion - No | 21 | 21 | 42
  Seminal Vesical Invasion -Yes | 3 | 0 | 3
Pelvic Lymph Node Dissection (PLND) [Count of Participants; unit: Participants]
  PLND - No | 5 | 5 | 10
  PLND -Yes | 19 | 16 | 35
weight of prostate [Mean (Standard Deviation); unit: grams] | 69.53 (35.92) | 54.30 (14.79) | 62.42 (28.66)
Operative time [Mean (Standard Deviation); unit: minutes] | 186.4 (54.6) | 171.4 (32.3) | 179.4 (45.7)

OUTCOME MEASURES:

1. Primary Outcome: Catheter Related Pain: Visual Analog Score Rating
Description: Catheter related pain was measured using a visual analog score rating mean post-operative pain on a scale from 1 (no pain) to 10 (worst possible pain). The lower the score the better the outcome.
Time Frame: post-op day 5-7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Catheter 16 French | Catheter 20 French
Number analyzed (Participants) | 24 | 21
score on a scale | 2.67 (1.61) | 2.67 (1.68)

2. Secondary Outcome: Urinary Symptoms
Description: The International Prostate Symptom Score (I-PSS) is based on the answers to seven questions concerning urinary symptoms and one question concerning quality of life. Each question concerning urinary symptoms allows the patient to choose one out of six answers indicating increasing severity of the particular symptom. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic).The lower the score the better the outcome.
Time Frame: week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Catheter 16 French | Catheter 20 French
Number analyzed (Participants) | 24 | 21
score on a scale | 9.81 (4.25) | 7.95 (4.04)

3. Secondary Outcome: Quality of Life Score
Description: Question eight of IPSS refers to the patient's perceived quality of life. The range is from delighted with a score of zero to terrible with a score of 6. The lower the score the better the outcome.
Time Frame: Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Catheter 16 French | Catheter 20 French
Number analyzed (Participants) | 24 | 21
score on a scale | 3 (1.3) | 2.95 (1.72)

4. Secondary Outcome: Urinary Symptoms
Description: The International Prostate Symptom Score (I-PSS) is based on the answers to seven questions concerning urinary symptoms and one question concerning quality of life. Each question concerning urinary symptoms allows the patient to choose one out of six answers indicating increasing severity of the particular symptom. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic).The lower the score the better the outcome.
  Question eight refers to the patient's perceived quality of life. The range is from delighted with a score of zero to terrible with a score of 6. The lower the score the better the outcome.
Time Frame: week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Catheter 16 French | Catheter 20 French
Number analyzed (Participants) | 24 | 21
score on a scale | 6.52 (4.75) | 7.59 (4.39)

5. Secondary Outcome: Quality of Life Score
Description: Question eight of the International Prostate Symptom Score (IPSS) refers to the patient's perceived quality of life. The range is from delighted with a score of zero to terrible with a score of 6. The lower the score the better the outcome
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Catheter 16 French | Catheter 20 French
Number analyzed (Participants) | 24 | 21
score on a scale | 2.24 (1.3) | 2.29 (1.05)

6. Secondary Outcome: Opioid Use
Description: Patient reported use of the number of tablets taken from provided prescription of opioids for post-operative pain. This will be converted to a standardized morphine equivalency for comparison. The lower the value the better the outcome.
Time Frame: after discharge until post-op day 7
Measure: Mean (Standard Deviation); unit: tablets
Arm/Group | Catheter 16 French | Catheter 20 French
Number analyzed (Participants) | 24 | 21
tablets | 5.00 (5.68) | 4.48 (5.75)

7. Secondary Outcome: Home Opioid Use in Standard Morphine Equivalency
Description: as for outcome 6
Time Frame: after discharge until post-op day 7
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Catheter 16 French | Catheter 20 French
Number analyzed (Participants) | 24 | 21
milligrams | 37.50 (42.60) | 33.57 (43.12)

8. Secondary Outcome: Number of Incontinence Pads Used
Description: Patient reported number of incontinence pads used per day. The lower the number the better the outcome.
Time Frame: week 6
Measure: Mean (Standard Deviation); unit: number of pads
Arm/Group | Catheter 16 French | Catheter 20 French
Number analyzed (Participants) | 24 | 21
number of pads | 2.00 (1.50) | 1.79 (1.32)

9. Secondary Outcome: Patient Reported Number of Pads Used Per Day.
Description: Patient reported number of incontinence pads used per day. The lower the number the better the outcome.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: number of pads
Arm/Group | Catheter 16 French | Catheter 20 French
Number analyzed (Participants) | 24 | 21
number of pads | 1.17 (1.46) | 1.13 (0.96)

10. Secondary Outcome: Number of Participants Experiencing Bladder Neck Contracture
Description: Number of incidence of participants experiencing bladder neck contracture.
Time Frame: week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Catheter 16 French | Catheter 20 French
Number analyzed (Participants) | 24 | 21
Participants | 0 | 0

11. Secondary Outcome: Number of Participants Experiencing Bladder Neck Contracture
Description: Number of Incidence of participants experiencing bladder neck contracture.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Catheter 16 French | Catheter 20 French
Number analyzed (Participants) | 24 | 21
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Catheter 16 French | Catheter 20 French
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/21
Other Adverse Events (participants affected / at risk) | 0/24 | 1/21
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Catheter 16 French (N=24) | Catheter 20 French (N=21)
bladder neck contracture (Renal and urinary disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/09/NCT04098809/Prot_SAP_000.pdf